CLINICAL TRIAL: NCT04364139
Title: African American Study of Kidney Disease and Hypertension
Acronym: AASK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: AASK U01DK048648; U01DK048648 (NIH)
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Hypertensive Nephrosclerosis; Chronic Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Ramipril; Amlodipine; Metoprolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants and investigators were masked to randomized drug but not BP goal
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Lower BP goal and Ramipril (Experimental): Participants assigned to Lower Blood Pressure Goal (MAP less than or equal to 92 mm Hg) and Participants assigned to Receive Ramipril 2.5 to 10 mg/d
  Interventions: Other: MAP goal less than or equal to 92 mm Hg; Drug: Ramipril
- Usual BP goal and Ramipril (Experimental): Participants assigned to usual Blood Pressure Goal (MAP of 102 to 107 mm Hg) and participants assigned to Receive Ramipril 2.5 to 10 mg/d
  Interventions: Other: MAP goal 102-107 mm Hg; Drug: Ramipril
- Lower BP goal and Amlodipine (Experimental): Participants assigned to Lower Blood Pressure Goal (MAP less than or equal to 92 mm Hg) and Participants assigned to Receive Amlodipine 5 to 10 mg/d
  Interventions: Other: MAP goal less than or equal to 92 mm Hg; Drug: Amlodipine
- Usual BP goal and Amlodipine (Experimental): Participants assigned to usual Blood Pressure Goal (MAP of 102 to 107 mm Hg) and Participants assigned to Receive Amlodipine 5 to 10 mg/d
  Interventions: Other: MAP goal 102-107 mm Hg; Drug: Amlodipine
- Lower BP goal and Metoprolol (Experimental): Participants assigned to Lower Blood Pressure Goal (MAP less than or equal to 92 mm Hg) and Participants assigned to Receive Metoprolol 50 to 200 mg/d
  Interventions: Other: MAP goal less than or equal to 92 mm Hg; Drug: Metoprolol
- Usual BP goal and Metoprolol (Experimental): Participants assigned to usual Blood Pressure Goal (MAP of 102 to 107 mm Hg) and Participants assigned to Receive Metoprolol 50 to 200 mg/d
  Interventions: Other: MAP goal 102-107 mm Hg; Drug: Metoprolol

INTERVENTIONS:
Other: MAP goal less than or equal to 92 mm Hg — Lower Blood Pressure Goal (mean arterial pressure (MAP) less than or equal to 92 mm Hg) which corresponds to a BP of approximately 115/80 mmHg
  Arms: Lower BP goal and Amlodipine; Lower BP goal and Metoprolol; Lower BP goal and Ramipril
Other: MAP goal 102-107 mm Hg — Usual Blood Pressure Goal (mean arterial pressure (MAP) 102-107 mm Hg) which corresponds to a BP of approximately 135/85 to 140/90 mmHg
  Arms: Usual BP goal and Amlodipine; Usual BP goal and Metoprolol; Usual BP goal and Ramipril
Drug: Ramipril — An angiotensin-converting enzyme inhibitor, (ACEI: ramipril) 2.5 to 10 mg/d
  Other Names: ACEI
  Arms: Lower BP goal and Ramipril; Usual BP goal and Ramipril
Drug: Amlodipine — A dihydropyridine calcium channel blocker, (DHPCCB: amlodipine) 5 to 10 mg/d
  Other Names: DHPCCB
  Arms: Lower BP goal and Amlodipine; Usual BP goal and Amlodipine
Drug: Metoprolol — A sustained release beta-blocker, (BB: metoprolol) 50 to 200 mg/d
  Other Names: BB
  Arms: Lower BP goal and Metoprolol; Usual BP goal and Metoprolol

SUMMARY:
The AASK is a multicenter, randomized, controlled clinical trial using a 2 × 3 factorial design to evaluate the effects of level of blood pressure control and type of anti-hypertensive medication on progression of chronic renal disease among African American men and women with chronic renal insufficiency caused by hypertension (hypertensive nephrosclerosis).

DETAILED DESCRIPTION:
The AASK is a multicenter, randomized, controlled clinical trial using a 2 × 3 factorial design to evaluate the effects of level of blood pressure control and type of anti-hypertensive medication on progression of chronic renal disease among African American men and women with chronic renal insufficiency caused by hypertension (hypertensive nephrosclerosis). Two levels of blood pressure control were defined in terms of mean arterial pressure (MAP = 2/3 diastolic blood pressure + 1/3 systolic blood pressure). A usual goal is defined as an MAP of 102 to 107 mm Hg, and a low goal is defined as an MAP of 92 mm Hg or less. The three antihypertensive drug regimens contained either a calcium channel blocker (amlodipine), β-blocker (metoprolol; Toprol XL), or angiotensin-converting enzyme inhibitor (ramipril) as initial therapy. Progression of renal disease was measured as the rate of decline in glomerular filtration rate (GFR).

ELIGIBILITY:
Inclusion Criteria:

1. African-American men and women (including black individuals born in the Caribbean, Africa, Canada, etc.) age 18 to 70 years. Each center will attempt to include equal numbers of men and women, at least 1:3 of each.
2. Hypertension is defined as a sitting diastolic BP of 95 mmHg or more. The average of the last two of three consecutive readings on a random zero sphygmomanometer machine at any visit is the level used. Hypertensive participants on anti-hypertensive therapy at Baseline need only one qualifying clinic visit. Those not currently on medications at Baseline must qualify on each of two consecutive clinic visits.
3. Reduced renal function, defined as a prerandomization (G1 visit) 125I-iothalamate GFR between 20 to 65 ml/min 1.73 per m^2.
4. Willingness and ability to cooperate with the protocol.

Exclusion Criteria:

1. History of malignant or accelerated hypertension within 6 mo prior to study entry; previous chronic peritoneal or hemodialysis or renal transplantation.
2. Known secondary causes of hypertension.
3. Any known history of diabetes mellitus type I and II, or fasting (8-12 h) glucose >140 mg/dl on two occasions, or glucose >200 mg/dl on one occasion prior to randomization.
4. A ratio of urinary protein (mg/dl) to creatinine (mg/dl) exceeding 2.5 in a 24-h urine sample collected shortly before the initial GFR visit. (This ratio is used as an estimate of > 2.5 g/d proteinuria without needing to factor for validity of the collection.)
5. Clinical or renal biopsy evidence of any renal disease other than hypertensive nephrosclerosis. Persons with arteriographically documented renal arterial atherosclerotic disease less than 50% stenosis of the renal artery should be considered eligible for study participation if the principal investigator at the center feels the disease is not clinically significant.
6. History of drug abuse in the past 2 yr, including narcotics, cocaine, or alcohol (>21 drinks/wk).
7. Serious systemic disease that might influence survival or the course of renal disease. (Chronic oral steroid therapy is an exclusion, but steroid-containing nasal sprays are not. In active sarcoidosis is not an exclusion.)
8. Clinical evidence of lead intoxication.
9. Arm circumference >52 cm, which precludes measuring blood pressure with the "thigh" blood pressure cuff. Arm length such that if the cuff that is appropriate for the arm circumference extends into the antecubital space so that the cuff would interfere with placement of the stethoscope over the brachial artery for blood pressure measurement.
10. Clinical evidence of congestive heart failure, current or within the preceding 6 mn. Ejection fraction below 35% measured by any method. Heart block greater than first degree or any other arrhythmia that would contraindicate the use of any of the randomized drugs.
11. Reactive airway disease, current or in the preceding 6 mo requiring prescribed treatment for more than 2 wk.
12. Impairment or difficulty in voiding, precluding adequate urine collections.
13. Intake of nonsteroidal anti-inflammatory agents (NSAIDs) more than 15 d/mo, excluding aspirin. Inability to discontinue NSAIDs or aspirin for 5 d prior to GFR measurement.
14. History of severe adverse reaction to any of the randomized drugs required for use in the protocol or contraindication of their use.
15. Pregnancy or likelihood of becoming pregnant during the study period; lactation.
16. Serum potassium level >5.5 mEq/L at the study visit 2 (SV2) and confirmed at G1 for those not on ACE inhibitors during baseline, or serum potassium level >5.9 mEq/L at the SV2 and confirmed at G1 for those on ACE inhibitors during baseline.
17. Leukopenia <2,500/mm3 at SV2 and confirmed at the end of baseline.
18. Medically indicated need for any of the randomized drugs for any other reason (including angina pectoris, migraine, arrhythmia).
19. Allergy to iodine.
20. Suspicion that the participant will not be able to adhere to medications or comply with the protocol visit schedule.
21. Participation in another intervention study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1094 (Actual)
Dates: Start 1995-02-01 (Actual); Primary Completion 2001-09-30 (Actual); Study Completion 2007-06-30 (Actual)

PRIMARY OUTCOMES:
Rate of change in GFR | Up to 3 years
  GFR slope was determined separately during the first 3 months after randomization (acute phase) and during the remainder of follow-up (chronic phase)

SECONDARY OUTCOMES:
Time to 50% reduction in GFR, ESRD, or death up to 3 years | Up to 3 years
  Time from randomization to any of the following (1) confirmed reduction in GFR by 50% or by 25 mL/min per 1.73 m^2, (2) end stage renal disease (ESRD), or (3) death
Change in proteinuria | Baseline to 3 years
  Change in proteinuria from baseline to the end of follow-up
Time to 50% reduction in GFR, ESRD, or death up to 10 years | Up to 10 years
  Time from randomization to any of the following (1) confirmed reduction in GFR by 50% or by 25 mL/min per 1.73 m^2, (2) end stage renal disease (ESRD), or (3) death

CONTACTS AND LOCATIONS:
Overall Officials: JENNIFER GASSMAN, Principal Investigator — CLEVELAND CLINIC LERNER COM-CWRU

IPD SHARING:
Plan to Share IPD: Yes
Data and samples are available at the National Institute of Diabetes Digestive and Kidney Diseases (NIDDK) Central Repository
Supporting Information: Study Protocol, CSR, Analytic Code
URL: https://repository.niddk.nih.gov/studies/aask-trial/?query=aask

REFERENCES:
- [Result] Agodoa LY, Appel L, Bakris GL, Beck G, Bourgoignie J, Briggs JP, Charleston J, Cheek D, Cleveland W, Douglas JG, Douglas M, Dowie D, Faulkner M, Gabriel A, Gassman J, Greene T, Hall Y, Hebert L, Hiremath L, Jamerson K, Johnson CJ, Kopple J, Kusek J, Lash J, Lea J, Lewis JB, Lipkowitz M, Massry S, Middleton J, Miller ER 3rd, Norris K, O'Connor D, Ojo A, Phillips RA, Pogue V, Rahman M, Randall OS, Rostand S, Schulman G, Smith W, Thornley-Brown D, Tisher CC, Toto RD, Wright JT Jr, Xu S; African American Study of Kidney Disease and Hypertension (AASK) Study Group. Effect of ramipril vs amlodipine on renal outcomes in hypertensive nephrosclerosis: a randomized controlled trial. JAMA. 2001 Jun 6;285(21):2719-28. doi: 10.1001/jama.285.21.2719. PMID 11386927
- [Result] Appel LJ, Wright JT Jr, Greene T, Agodoa LY, Astor BC, Bakris GL, Cleveland WH, Charleston J, Contreras G, Faulkner ML, Gabbai FB, Gassman JJ, Hebert LA, Jamerson KA, Kopple JD, Kusek JW, Lash JP, Lea JP, Lewis JB, Lipkowitz MS, Massry SG, Miller ER, Norris K, Phillips RA, Pogue VA, Randall OS, Rostand SG, Smogorzewski MJ, Toto RD, Wang X; AASK Collaborative Research Group. Intensive blood-pressure control in hypertensive chronic kidney disease. N Engl J Med. 2010 Sep 2;363(10):918-29. doi: 10.1056/NEJMoa0910975. PMID 20818902
- [Result] Wright JT Jr, Bakris G, Greene T, Agodoa LY, Appel LJ, Charleston J, Cheek D, Douglas-Baltimore JG, Gassman J, Glassock R, Hebert L, Jamerson K, Lewis J, Phillips RA, Toto RD, Middleton JP, Rostand SG; African American Study of Kidney Disease and Hypertension Study Group. Effect of blood pressure lowering and antihypertensive drug class on progression of hypertensive kidney disease: results from the AASK trial. JAMA. 2002 Nov 20;288(19):2421-31. doi: 10.1001/jama.288.19.2421. PMID 12435255